CLINICAL TRIAL: NCT07274046
Title: Clinical and Public-Health Impact of Tick-Borne Encephalitis: A Prospective Multicenter Observational Study With 12-Month Follow-up and Cost-Effectiveness Analysis
Brief Title: Burden of Tick-borne Encephalitis and Cost-effectiveness of Vaccination in the Czech Republic
Acronym: ENCZECH
Status: Recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: České Budějovice Hospital (Other); University Hospital Ostrava (Other); Hospital Pardubice (Unknown); Bulovka Hospital (Other)
Responsible Party: Principal Investigator, Martin Slížek, Principal Investigator, Department of Infectious Diseases, Charles University, Czech Republic
Other Study IDs: TBE-CZ-OBS-2023-01; 06_SM_FNB_002 (Other Grant/Funding Number: Bulovka University Hospital)
Record Dates: First submitted 2025-11-19; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Tick Borne Encephalitis (TBE)
Keywords: tick-borne encephalitis; sequelae; post-encephalitic syndrome; age; TBEV; encephalitis; cost-effectiveness
MeSH Terms: conditions — Encephalitis, Tick-Borne; Encephalitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TBE cohort: Children and adults hospitalized with confirmed tick-borne encephalitis, followed prospectively for 12 months.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational study only. Participants receive standard clinical care; no experimental or study-specific interventions are administered.

SUMMARY:
This observational study follows children and adults who were hospitalized with tick-borne encephalitis (TBE) in the Czech Republic. The aim is to better understand how individuals recover from TBE, which symptoms may persist after the infection, and which patients may require additional support during their recovery. Participants are examined several times after hospital discharge (at 2-4 weeks, 3 months, 6 months, and 12 months) to observe changes in symptoms, functional status, and daily activities. Follow-up assessments include evaluation of common post-infection problems such as tiredness, headaches, memory or concentration difficulties, sleep issues, or limb weakness. Symptoms lasting for several months are categorized as post-encephalitic syndrome (PES).

The study also assesses how TBE affects daily functioning, school and work performance, and overall quality of life using questionnaires and short functional assessments. In addition, the study includes a public-health component that estimates the broader impact of TBE in the population and evaluates the potential benefits of vaccination in preventing long-term health complications.

The findings aim to support improved patient care, follow-up planning, and evidence-based public-health decision-making in the Czech Republic.

DETAILED DESCRIPTION:
Tick-borne encephalitis (TBE) is a serious viral infection of the central nervous system and represents a longstanding public-health challenge in the Czech Republic, a country with one of the highest TBE incidences in Europe. Although an effective vaccine has been available for decades, population-level vaccination coverage remains low, resulting in persistently high incidence across all age groups and numerous severe cases requiring hospitalization. Despite extensive clinical experience with TBE, the long-term course of the disease, the full spectrum of postencephalitic syndrome (PES), and the associated functional and neurocognitive burden remain incompletely quantified in contemporary, real-world populations. Updated evidence is also needed to inform public-health planning and to evaluate the potential health and economic benefits of broader TBE vaccination in this high-endemicity setting.

The study is a prospective multicenter observational investigation enrolling children and adults hospitalized with laboratory-confirmed TBE across four major infectious disease centers in the Czech Republic. Standardized clinical and functional assessments are applied to capture both the acute clinical course and the long-term recovery trajectory. Acute disease severity is classified using predefined clinical criteria, including the presence of motor deficit (paresis) during hospitalization, intensive-care unit admission, prolonged hospitalization (length of stay >10 days), or death. Follow-up assessments occur at 2-4 weeks, 3 months, 6 months, and 12 months after discharge.

Long-term outcomes are evaluated using validated tools, including the modified Rankin Scale (mRankin) to assess global functional disability and the Minimum European Health Module (MEHM) to capture self-perceived health, activity limitation, and chronic morbidity. A central focus of the study is the characterization of postencephalitic syndrome (PES), the most common long-term complication of TBE. PES is defined as the persistence of one or more neurological, cognitive, or functional symptoms lasting for at least 6 months after acute infection. These symptoms may include chronic fatigue, impaired concentration or memory, cognitive slowing, sleep disturbances, headaches, irritability, anxiety, or reduced exercise tolerance. Persistent motor deficits, such as paresis or impaired coordination, are evaluated as integral components of PES, reflecting a more severe neurological phenotype. Detailed symptom-level data and functional assessments are collected to comprehensively describe the prevalence, severity, and heterogeneity of PES and its impact on long-term quality of life.

The study examines demographic and clinical predictors of adverse outcomes, including the role of age, comorbidities, markers of central nervous system involvement during the acute phase, and initial disease severity. These analyses are intended to support improved prognostic counseling and inform follow-up and rehabilitation strategies.

A public-health and economic component quantifies the overall burden of TBE in disability-adjusted life years (DALYs), integrating observed functional outcomes, sequelae duration, disability weights, and TBE-related mortality. DALY estimates are combined with national epidemiological surveillance data to ensure representativeness across age groups and regions. These outcomes will form the basis for a decision-analytic model evaluating the cost-effectiveness of increasing TBE vaccination coverage. The model compares current vaccination uptake with expanded coverage scenarios across different age groups and generates estimates of incremental cost-effectiveness ratios (ICERs), projected health gains, reductions in long-term disability, and potential healthcare cost savings. The economic modeling relies solely on aggregated clinical and epidemiological data and does not include any patient-level interventions.

By integrating prospective clinical follow-up, standardized functional assessments, detailed characterization of PES, and health-economic modeling, the study provides a comprehensive evaluation of the clinical and economic burden of TBE in the Czech Republic. The findings may inform clinical practice, long-term patient management, and national vaccination policy, contributing to improved prevention and mitigation of TBE-related morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization due to suspected central nervous system (CNS) infection.
* Laboratory-confirmed TBE, defined as:

the presence of CNS symptoms and cerebrospinal fluid pleocytosis (>5 × 10⁶/L) and TBEV IgM and IgG seropositivity in serum, or detection of TBEV IgM in CSF in previously vaccinated individuals.

* All age groups (children and adults).
* Ability to participate in scheduled follow-up (in person or via telephone).
* Informed consent provided by the patient or legal guardian (for minors).

Exclusion Criteria:

* Alternative diagnosis explaining the CNS symptoms
* Missing essential clinical or laboratory data required to confirm TBE or assess outcomes.
* Refusal or inability to provide informed consent.
* Inability to complete follow-up assessments, including situations where reliable contact cannot be maintained.
* Coexisting severe neurological disorder unrelated to TBE that prevents meaningful evaluation of sequelae (e.g., advanced neurodegenerative disease, severe preexisting motor disability).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized children and adults with confirmed tick-borne encephalitis (TBE) treated at four infectious disease centers in the Czech Republic. All participants had clinical symptoms of central nervous system involvement, cerebrospinal fluid pleocytosis, and laboratory confirmation of TBEV infection. Patients were enrolled during their acute hospitalization and followed prospectively for up to 12 months as part of a standardized clinical and functional outcome assessment program.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Presence and Severity of Post-Encephalitic Syndrome (PES) | 6 months post-discharge and 12 months post-discharge
  PES is defined as the presence of ≥1 neurological, cognitive, or functional symptom persisting ≥6 months after acute TBE. PES severity is graded as:
  Mild: mRankin = 1, no limitation of usual activities Moderate: mRankin = 2 and/or limited but preserved independence, or poor self-perceived health (MEHM) Severe: mRankin ≥3, severe limitation of daily activities, very poor self-perceived health, or death.

SECONDARY OUTCOMES:
Persistent Motor Deficit | 6 months post-discharge and 12 months post-discharge
  Presence of persistent paresis or other objective motor impairment at follow-up attributed to TBE.
Acute Disease Severity Classification | During index hospitalization
  Acute course categorized as severe if any of the following criteria are present:
  motor deficit (paresis) during hospitalization, ICU admission, hospitalization >10 days, death. All others classified as mild.
Functional Status by Modified Rankin Scale (mRankin) | 2-4 weeks post-discharge; 3 months; 6 months; 12 months
  Global functional disability assessed by mRankin (0-6).
Self-perceived Health and Activity Limitation (MEHM Score) | 2-4 weeks post-discharge; 3 months; 6 months; 12 months
  Minimum European Health Module (MEHM), including perceived health, activity limitation, and chronic morbidity.
Persistence or Resolution of Individual PES Symptoms (Structured Symptom Checklist) | 2-4 weeks post-discharge; 3 months; 6 months; 12 months
  This outcome is assessed using a structured PES Symptom Checklist developed for standardized evaluation of post-encephalitic symptoms. The checklist captures the presence or absence of individual symptoms associated with post-encephalitic syndrome (PES), including fatigue, exertion intolerance, headache, cognitive slowing, memory problems, concentration difficulties, sleep disturbances, sensory deficits, and emotional instability.
  Each symptom is recorded as present or absent at each follow-up assessment.
  The outcome will be reported as:
  number of symptoms present (range 0-X), and presence/absence of each individual symptom (binary assessment).
  Unit of Measure:
  Number of symptoms (count) and binary presence/absence for each symptom
Hospital Length of Stay (LOS) | From hospital admission to hospital discharge, assessed over an expected hospitalization period of up to 90 days.
  Total duration of the index hospital stay in days, from hospital admission for acute TBE to hospital discharge.
ICU Admission | From hospital admission to hospital discharge, including any ICU stay, assessed over an expected hospitalization period of up to 90 days.
  Whether the patient was admitted to intensive care during acute TBE and the length of ICU stay.
All-Cause Mortality (binary outcome) | During index hospitalization; 6 months post-discharge; 12 months post-discharge
  All-cause mortality recorded as a binary outcome (alive/deceased) at predefined time points. Mortality during the index hospitalization and mortality during follow-up (6 and 12 months post-discharge) are recorded separately.
  Unit of Measure: Proportion of participants deceased (%)
Cost-Effectiveness of TBE Vaccination | Final analysis at 12 months after completion of follow-up.
  Cost-effectiveness of increasing TBE vaccination coverage in the Czech Republic based on disability-adjusted life years (DALYs) derived from observed functional outcomes (mRankin, MEHM), PES prevalence, symptom duration, and TBE-associated mortality. A decision-analytic model will estimate incremental cost-effectiveness ratios (ICERs) across different age groups and vaccination coverage scenarios using real-world clinical data combined with national surveillance data.
Change in Functional Status (modified Rankin Scale, mRankin) | Baseline (hospitalization), 2-4 weeks post-discharge, 3 months, 6 months, 12 months.
  Change in global functional disability assessed using the modified Rankin Scale (0-6). Scores are recorded at each follow-up visit to evaluate recovery trajectory and functional outcomes after acute TBE.
Change in Self-Perceived Health (Minimum European Health Module, MEHM) | Baseline (hospitalization), 2-4 weeks post-discharge, 3 months, 6 months, 12 months.
  Change in self-perceived health, activity limitation, and chronic morbidity assessed using the Minimum European Health Module (MEHM).
  Unit of Measure: MEHM score (categorical responses)

CONTACTS AND LOCATIONS:
Locations (4):
- Czechia (4):
  - České Budějovice Hospital, České Budějovice, Jihočeský kraj
  - Ostrava University Hospital, Ostrava, Moravskoslezský kraj
  - Pardubická nemocnice, Pardubice, Pardubický kraj
  - Bulovka University Hospital, Prague, Prague

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Only aggregated, anonymized results will be made available in publications.